CLINICAL TRIAL: NCT00531245
Title: A Phase I/II Trial of TS-1 and Oxaliplatin in Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Young Suk Park, Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-01-024
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2007-08

CONDITIONS: Colorectal Neoplasms
Keywords: TS-1 and oxaliplatin; Phase I/II study; Colorectal cancer; First line treatment
MeSH Terms: conditions — Colorectal Neoplasms | interventions — titanium silicide; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: TS-1, oxaliplatin — Oxaliplatin(130 mg/m2) day 1, intravenously TS-1 at a dose of 60, 70, 80, 90, 100, 110, 120 mg/m2 given orally starting day 1 until day 14(2 weeks ON, 1 weeks OFF), every 3 weeks

SUMMARY:
Capecitabine and oxaliplatin(XELOX) is active first-line therapy for patients with metastatic colorectal cancer. Phase II study of TS-1, a novel oral fluoropyrimidine derivative, showed activity in patients with metastatic colorectal carcinoma. Preclinical data of TS-1 with oxaliplatin showed synergistic activity in vivo human colorectal cancer xenograft. There is no data about the optimal dose of TS-1 with 2 weeks schedule combined with oxaliplatin. Therefore in a phase I study, we would like to determine the maximum tolerated dose(MTD) of TS-1 and oxaliplatin and define the recommended dose for subsequent phase II study. And then, in a phase II study we would like to evaluate the efficacy(response rates) and toxicities of the new combination regimen in advanced colorectal cancer.

DETAILED DESCRIPTION:
Subjects meeting all of the following criteria will be considered for enrolment into the study.

1. Histologically documented colorectal adenocarcinoma
2. Previous chemotherapy up to two regimens(including adjuvant chemotherapy and first-line chemotherapy without oxaliplatin) is allowed in phase I portion; patients are required to have discontinued chemotherapy and/or radiotherapy for at least 4weeks before entry into phase I portion. No prior chemotherapy or radiotherapy allowed(adjuvant chemotherapy and/or radiotherapy would be allowed) in phase II portion
3. Age 18 to 75 years old
4. At least one unidimensional measurable lesion with a diameter >20 mm using conventional CT or MRI scans or >10 mm using spiral CT scans (use of spiral CT must be documented in medical records and used consistently throughout study).
5. In phase I study, prior radiotherapy is permitted if it was not administered to target lesions selected for this study, unless progression of the selected target lesions within the radiation portal is documented, and provided it has been completed at least 4 weeks before study entry.
6. Performance status (ECOG scale): 0-2
7. Patients can take food and drugs orally
8. Adequate organ functions
9. Life expectancy ≥ 3 months
10. Written informed consent

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented colorectal adenocarcinoma
* Previous chemotherapy up to two regimens(including adjuvant chemotherapy and first-line chemotherapy without oxaliplatin) is allowed in phase I portion; patients are required to have discontinued chemotherapy and/or radiotherapy for at least 4weeks before entry into phase I portion. No prior chemotherapy or radiotherapy allowed(adjuvant chemotherapy and/or radiotherapy would be allowed) in phase II portion
* Age 18 to 75 years old
* At least one unidimensional measurable lesion using spiral CT scans (use of spiral CT must be documented in medical records and used consistently throughout study).
* In phase I study, prior radiotherapy is permitted if it was not administered to target lesions selected for this study, unless progression of the selected target lesions within the radiation portal is documented, and provided it has been completed at least 4 weeks before study entry.
* Performance status (ECOG scale): 0-2
* Patients can take food and drugs orally
* Adequate organ functions
* Life expectancy more than 3 months
* Written informed consent

Exclusion Criteria:

* Tumor type other than adenocarcinoma
* Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or prior malignancy treated more than 5 years ago without recurrence)
* Prior chemotherapy with TS-1 and/or oxaliplatin
* Presence of CNS metastasis
* Obvious peritoneal seeding or bowel obstruction disturbing oral intake
* Evidence of serious gastrointestinal bleeding requiring transfusion
* Symptomatic peripheral neuropathy (NCI CTC v3.0 greater than Grade I)
* Major surgery within 4 weeks prior to study treatment start, or lack of complete recovery from the effects of major surgery.
* Serious illness or medical conditions, as follows; uncontrolled congestive heart failure, angina pectoris, arrhythmias, or hypertension, hepatic cirrhosis, interstitial pneumonia, pulmonary adenomatosis, psychiatric disorder that may interfere with and/or protocol compliance, unstable diabetes mellitus, uncontrolled ascites or pleural effusion, active infection
* Pregnant or lactating woman
* Women of child bearing potential not using a contraceptive method
* Receiving a concomitant treatment with drugs interacting with TS-1 or oxaliplatin, as follows; flucytosine, a fluorinated pyrimidine antifungal agent, phenytoin, warfarin
* Received any investigational drug or agent/procedure, i.e. participation in another trial within 4 weeks before beginning treatment with study drug.
* Any patients judged by the investigator to be unfit to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2006-08; Primary Completion 2008-06 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
In a phase I study, to determine the maximum tolerated dose(MTD) In a phase II study, to evaluate the efficacy(response rates) and toxicities | one year

SECONDARY OUTCOMES:
To investigate the time to progression(TTP), overall survival and toxicity | two year

CONTACTS AND LOCATIONS:
Overall Officials: Young Suk Park, M.D., Ph.D., Principal Investigator — Samsung Medical Center, Seoul, KOREA
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Naktsuka M, Saito H, et al., A new combination chemotherapy based on oral fluoropyrimidine, TS-1 combined with oxaliplatin is highly effective against colorectal cancer in vivo 97th AACR Annual Meeting, #4730, 2006
- [Result] Cassidy J, Tabernero J, Twelves C, Brunet R, Butts C, Conroy T, Debraud F, Figer A, Grossmann J, Sawada N, Schoffski P, Sobrero A, Van Cutsem E, Diaz-Rubio E. XELOX (capecitabine plus oxaliplatin): active first-line therapy for patients with metastatic colorectal cancer. J Clin Oncol. 2004 Jun 1;22(11):2084-91. doi: 10.1200/JCO.2004.11.069. PMID 15169795
- [Result] Shirao K, Ohtsu A, Takada H, Mitachi Y, Hirakawa K, Horikoshi N, Okamura T, Hirata K, Saitoh S, Isomoto H, Satoh A. Phase II study of oral S-1 for treatment of metastatic colorectal carcinoma. Cancer. 2004 Jun 1;100(11):2355-61. doi: 10.1002/cncr.20277. PMID 15160338
- [Result] Emura T, Suzuki N, Yamaguchi M, Ohshimo H, Fukushima M. A novel combination antimetabolite, TAS-102, exhibits antitumor activity in FU-resistant human cancer cells through a mechanism involving FTD incorporation in DNA. Int J Oncol. 2004 Sep;25(3):571-8. PMID 15289858